CLINICAL TRIAL: NCT01935570
Title: Comparative Study of the Bioavailability of Magnesium Administrated by Two ChronoMag Smart Tablet® 50 mg Versus Three Mag2® Tablets 100mg.
Acronym: BioChronoMag
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr Gisèle PICKERING (MCU-PH)(Clinical Pharmacology center, Inserm 501) (Unknown); Dr Gilles DUCHEIX (Attaché)(Clinical Pharmacology center, Inserm 501) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0162
Record Dates: First submitted 2013-07-02; First posted 2013-09-05 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
Keywords: Bioavailability of magnesium; Digestive and general tolerance
MeSH Terms: interventions — Magnesium Chloride; magnesium carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Magnesium (Experimental)
  Interventions: Drug: Magnesium chloride (ChronoMag Smart Tablet®); Drug: Magnesium carbonate (Mag2® Tablet)

INTERVENTIONS:
Drug: Magnesium chloride (ChronoMag Smart Tablet®)
Drug: Magnesium carbonate (Mag2® Tablet)

SUMMARY:
This clinical study is composed of two steps. The first step aims at validating the pharmacokinetic approach based on the magnesium concentration in erythrocyte and plasma.

According to these results and if this pharmacokinetic approach is validated, the second step will set up. The second phase aims at comparing the relative bioavailability of magnesium administrated by two different drug formulations: ChronoMag Smart Tablet® (two tablets50mg) versus Mag2® (three tablets100mg).

DETAILED DESCRIPTION:
" Go/no go " comparative biodisponibility study. Randomised, cross-over, controlled and double-blind, monocentric study in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Patient aged between 18 and 50
* Patient with a normal blood magnesium rate between 0.65 and 1.05 mmol/l
* Patient with vital signs values considered as normal by the investigator before drug administration
* Sufficient cooperation and understanding to comply with the requirements of study.
* Patient without medication during the 7 days preceding the inclusion
* Acceptance to give a written consent.
* Affiliation at system of French social security.
* Inscription or acceptation of inscription at national register of voluntaries participant at research.

Exclusion Criteria:

* Against magnesium-indication: hypersensitivity known at carbonate or magnesium chloride or at one of the excipients.
* Patient with medication or supplementation of magnesium
* Severe renal insufficiency with a creatine clearance ≤ 30ml/min
* Medical and chirurgical history considered as incompatible with the study
* A progressive pathology during the inclusion
* A consumption of more than 50g of dark chocolate per day
* An excessive alcohol consumption, an excessive tobacco consumption ( more than 10 cigarettes a day), an excessive tea, coffee or drink with caffeine consumption or drug addictions
* Patient who participated in another clinical trial located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial.
* Patient with cooperation and understanding insufficiency to comply with the requirements of protocol
* Minor or patient with social protection (curatorship, tutorship…)
* No affiliation at system of French social security

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
blood magnesium concentration | T0, T0+30 minutes, T0+1h, T0+2h, T0+3h, T0+4h, T0+5h, T0+6h, T0+7h, T0+8h).
urine magnesium concentration | T0+5h , T0+10h , T0+24h

SECONDARY OUTCOMES:
Adverse digestive events record | T0+24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christian DUALE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France